CLINICAL TRIAL: NCT07157969
Title: Immune Checkpoint Inhibitors and Anti-Vascular Endothelial Growth Factor Antibody/Tyrosine Kinase Inhibitors With or Without Interventional Therapy for Advanced HCC
Brief Title: ICIs and Anti-VEGF Antibody/TKIs With or Without Interventional Therapy for Advanced HCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K7470
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-02

CONDITIONS: HCC - Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib; pembrolizumab; atezolizumab; Bevacizumab; camrelizumab; apatinib; tislelizumab; sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immune checkpoint inhibitors combined with anti-VEGF drugs (Active Comparator): Immune checkpoint inhibitors include Pembrolizumab, Atezolizumab, Camrelizumab, Tislelizumab, and Sintilimab.
  Anti-VEGF drugs include Bevacizumab, Lenvatinib, and Apatinib.
  Interventions: Drug: Lenvatinib; Drug: Pembrolizumab; Drug: Atezolizumab; Drug: Bevacizumab; Drug: Camrelizumab; Drug: Apatinib; Drug: Tislelizumab; Drug: Sintilimab
- Immune checkpoint inhibitors combined with anti-VEGF drugs alongside interventional therapy (Experimental): Immune checkpoint inhibitors include Pembrolizumab, Atezolizumab, Camrelizumab, Tislelizumab, and Sintilimab.
  Anti-VEGF drugs include Bevacizumab, Lenvatinib, and Apatinib. Interventional therapy includes C-TACE, D-TACE, and HAIC.
  Interventions: Drug: Lenvatinib; Drug: Pembrolizumab; Drug: Atezolizumab; Drug: Bevacizumab; Drug: Camrelizumab; Drug: Apatinib; Procedure: TACE; Procedure: HAIC; Procedure: DEB-TACE; Drug: Tislelizumab; Drug: Sintilimab

INTERVENTIONS:
Drug: Lenvatinib — ≥60 kg: 12 mg once daily, or <60 kg: 8 mg once daily
Drug: Pembrolizumab — 200 mg intravenously every three weeks
Drug: Atezolizumab — 1200 mg intravenously every three weeks
Drug: Bevacizumab — 15mg/kg intravenously every three weeks
Drug: Camrelizumab — 200 mg intravenously every three weeks
Drug: Apatinib — 250mg once daily
Procedure: TACE — The specific number and interval of interventional therapy sessions will be determined according to the patient's individual condition.
  Arms: Immune checkpoint inhibitors combined with anti-VEGF drugs alongside interventional therapy
Procedure: HAIC — The specific number and interval of interventional therapy sessions will be determined according to the patient's individual condition.
  Arms: Immune checkpoint inhibitors combined with anti-VEGF drugs alongside interventional therapy
Procedure: DEB-TACE — The specific number and interval of interventional therapy sessions will be determined according to the patient's individual condition.
  Arms: Immune checkpoint inhibitors combined with anti-VEGF drugs alongside interventional therapy
Drug: Tislelizumab — 200 mg intravenously every three weeks
Drug: Sintilimab — 200 mg intravenously every three weeks

SUMMARY:
This trial is designed to explore the efficacy and safety of interventional therapy combined with immune checkpoint inhibitors(ICIs) and anti-vascular endothelial growth factor(VEGF) antibody/tyrosine kinase inhibitors in the treatment of advanced hepatocellular carcinoma. Eligible participants will be divided into two groups based on their treatment plans: one receiving ICIs combined with anti-VEGF drugs, and the other receiving ICIs combined with anti-VEGF drugs alongside interventional therapy, which includes C-TACE, D-TACE, and HAIC. The specific number and interval of interventional therapy sessions will be determined according to the patient's individual condition.

Researchers will closely monitor and rigorously evaluate the efficacy and safety of the treatment in participants through follow-up assessments. The primary endpoint is the objective response rate , while secondary endpoints include disease control rate, progression-free survival, overall survival, duration of response, adverse events, and serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participate in the study, provide written informed consent, demonstrate good compliance, and are cooperative with follow-up.
2. Age ≥18 years at the time of signing informed consent, regardless of gender.
3. Diagnosis of hepatocellular carcinoma confirmed by imaging (according to AASLD criteria), histology, or cytology.
4. BCLC Stage B or C.
5. At least one measurable lesion per RECIST 1.1.
6. ECOG score of 0-1.
7. Child-Pugh liver function class A or B.
8. Life expectancy ≥ 3 months.
9. Adequate hematological and organ function.

Exclusion Criteria:

1. Patients with hepatocellular carcinoma who are candidates for surgical radical cure, or have undergone radical surgery without evaluable lesions, or have a history of or are planned for liver transplantation.
2. Pregnant or breastfeeding women.
3. Individuals with known allergy or intolerance to recombinant humanized PD-1/PD-L1 monoclonal antibody preparations.
4. Received local-regional therapy within 4 weeks before the first dose of the study drug, including but not limited to surgery, radiotherapy, hepatic artery embolism, TACE, hepatic artery infusion, radiofrequency ablation, cryoablation, or percutaneous ethanol injection.
5. History of other malignant tumors within 5 years prior to screening, except for hepatocellular carcinoma.
6. Presence of unhealed severe wounds, active ulcers, or untreated fractures.
7. Active autoimmune disease or history of autoimmune disorders.
8. Significant history of gastrointestinal diseases.
9. Significant history of cardiovascular or cerebrovascular diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
ORR, objective response rate | 12 months after the last subject is enrolled

SECONDARY OUTCOMES:
PFS, progression free survival | 12 months after the last subject is enrolled
OS, overall survival | 12 months after the last subject is enrolled
DCR, disease control rate | 12 months after the last subject is enrolled
DoR, duration of response | 12 months after the last subject is enrolled
Adverse events (AE) | 12 months after the last subject is enrolled
Serious adverse events (SAE) | 12 months after the last subject is enrolled

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kudo M, Ren Z, Guo Y, Han G, Lin H, Zheng J, Ogasawara S, Kim JH, Zhao H, Li C, Madoff DC, Ghobrial RM, Kawaoka T, Gerolami R, Ikeda M, Kumada H, El-Khoueiry AB, Vogel A, Peng X, Mody K, Dutcus C, Dubrovsky L, Siegel AB, Finn RS, Llovet JM; LEAP-012 investigators. Transarterial chemoembolisation combined with lenvatinib plus pembrolizumab versus dual placebo for unresectable, non-metastatic hepatocellular carcinoma (LEAP-012): a multicentre, randomised, double-blind, phase 3 study. Lancet. 2025 Jan 18;405(10474):203-215. doi: 10.1016/S0140-6736(24)02575-3. Epub 2025 Jan 8. PMID 39798578